CLINICAL TRIAL: NCT06412718
Title: Validation of Human Drugs Target of Repurposed Drugs and Novel Therapies
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Giulio Ferrari, Professor of Ophthalmology-San Raffaele Vita Salute University, Cornea and Ocular Surface Unit; Head-Eye Repair Lab San Raffaele Scientific Institute, IRCCS Ospedale San Raffaele
Other Study IDs: RV-WP2
Record Dates: First submitted 2024-04-30; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Rare Diseases; Aniridia; Neurotrophic Keratopathy; Limbal Stem Cell Deficiency; Ocular Graft-versus-host Disease; Ocular Cicatricial Pemphigoid; EEC Syndrome; Corneal Neovascularization
Keywords: Rare Eye Diseases; Aniridia; Neurotrophic Keratopathy; Limbal Stem Cell Deficiency; Ocular Graft-versus-host Disease; Ocular Cicatricial Pemphigoid; Corneal Neovascularization; Molecular targets; Cellular targets; Genomic targets; NK1R; PBMC; Substance P; VEGF; Blood; Tear; Impression cytology; Cytokine
MeSH Terms: conditions — Rare Diseases; Aniridia; Limbal Stem Cell Deficiency; Pemphigoid, Benign Mucous Membrane; Ectrodactyly-cleft lip-palate syndrome; Corneal Neovascularization; Lacerations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients
- Control group

SUMMARY:
The cross-sectional observational clinical study related to rare eye diseases is a multi-center study in which the hypothesis is that neurokinin 1 receptor and/or substance P expression is increased in REDs associated with inflammation/pain. Moreover, the following alternative targets are: VEGF, PAX6 and pro-inflammatory cytokine.

The following procedures are performed specifically for the study: samples of blood, tear fluid and impression cytology.

Precisely during the ophthalmological exam performed according to normal clinical practice (uncorrected visual acuity, best spectacle corrected visual acuity, corneal topography, corneal pachymetry and the slit lamp pictures) investigator's team collect the samples of blood, tear fluid and impression cytology to evaluate the goal of the study.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for study group

* Women and men with age equal or higher than 18 years (patients in reproductive age may be included in the study).
* Willingness and ability to read and understand the informed consent.
* Diagnosis (including genotype, if needed) of REDs.

Inclusion Criteria for control group

* Women and men with age equal or higher than 18 years (patients in reproductive age may be included in the study).
* Willingness and ability to read and understand the informed consent.
* Non - diagnosis of REDs.

Exclusion Criteria:

Exclusion Criteria for study group

Patients who meet these criteria will be excluded from participation in the study:

* Pregnancy, breastfeeding.
* Active ocular infection.
* Descemetocele/impending corneal perforation.
* Recent (less than 3 months) ocular surgery.
* Recent (less than 1 month) change in topical medications type and frequency.

Exclusion Criteria for control group

Patients who meet these criteria will be excluded from participation in the study:

* Pregnancy, breastfeeding.
* Active ocular infection.
* Descemetocele/impending corneal perforation.
* Recent (less than 3 months) ocular surgery.
* Recent (less than 1 month) change in topical medications type and frequency.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of 137 patients, each of them will present with one of the 7 diseases under study (REDs).
  The control group will consist of 137 patients not presenting the previous reported REDs.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
To quantify the expression of molecular/cellular/genomic targets in the REDs and control group to detect statistically significant and clinically relevant differences. | Day 0 (enrollment day).
  Evaluation of NK1R transcription levels in PBMC, substance P and VEGF protein levels in the tear fluid, pro-inflammatory cytokines transcription levels in conjunctival tissue.
  NK1R and pro-inflammatory cytokines are expressed as fold change compared to control group.
  Substance P and VEGF are expressed as ng/ml.

SECONDARY OUTCOMES:
To correlate the expression of molecular/cellular genomic targets with the clinical phenotype/quality of life/pain symptoms in patients with the 7 rare diseases and in the control group so as to detect possible risk factors. | Day 0 (enrollment day).
  Levels of NK1R, substance P, VEGF, and pro-inflammatory cytokines correlated with pictures, questionnaires, uncorrected visual acuity, best spectacle corrected visual acuity, corneal topography, corneal pachymetry and the slit lamp pictures acquired during the ophthalmologic exam.

REFERENCES:
- See also: European Commission, ERN-EYE: a European Reference Network dedicated to Rare Eye Diseases. Accessed 29 December 2021 — https://www.ern-eye.eu/ern-eye-a-european-reference-network-dedicated-to-rare-eye-diseases/
- See also: European Blind Union, About Blindness and Partial Sight: Facts and Figures. Accessed 26 August 2022 — https://www.euroblind.org/about-blindness-and-partial-sight/facts-and-figures
- See also: Restore Vision site — https://restorevision-project.eu/